CLINICAL TRIAL: NCT02322203
Title: Evaluation of the Effects of Niacin Therapy on Lipoprotein Composition and Function
Brief Title: Effects of Niacin Therapy on Lipoprotein Composition and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 150042; 15-H-0042
Record Dates: First submitted 2014-12-20; First posted 2014-12-23 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
Keywords: Niacin; Cholesterol; High-Density Lipoprotein; Low-Density Lipoprotein; Lipoproteins
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Niacin

STUDY DESIGN:
Intervention Model Description: This novel pilot study will be carried out at the NIH Clinical Center outpatient clinic 7 in healthy volunteers. We will screen up to 200 subjects, males and females, to obtain at least 32 completed studies. Participants will be recruited via flyer, and/or recruitment advertisement placed in the NIH Record, the NHLBI Recruitment website, the Clinical Center News and by email/listserv.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niacin ER in healthy participants and its effects on lipoprotein composition and function (Experimental): Niacin extended release (ER) to be given as follows: 500 mg/day for 1 week, then 1000 mg/day for 1 week, then 2000 mg/day for 14 weeks in healthy participants.
  Interventions: Dietary Supplement: Niacin Extended Release

INTERVENTIONS:
Dietary Supplement: Niacin Extended Release — Subjects will receive a 2 week supply of the dietary supplement Rugby Extended Release Niacin (250 mg/tablet) Niacin and will be instructed to take 2 tablets per day (500 mg/day) for the first seven days and then increase to 4 tablets per day (1000 mg/day) during the following 7 days. Subjects will then be escalated to 2000 mg/day for 14 weeks.
  Other Names: Niacin Extended Release (ER); Niacin

SUMMARY:
Background:

- Niacin is a vitamin in many foods, including meats, fish, fruits, and vegetables. It is often used as a dietary supplement that causes many improvements in the body. Researchers think it can affect heart health.

Objective:

- To better understand the good effects of niacin supplementation on cholesterol, fat metabolism, and vascular health.

Eligibility:

- Adults 18 years of age and older with fasting good cholesterol (HDL-C) below 60 mg/dL.

Design:

* Participants will come to the clinic 4 times during the study.
* They will complete a 7-day food journal before visits 1 and 3.
* At visit 1, participants will be screened with questions about their diet and exercise, medical history, and any drugs and vitamins they take. Vital signs and body mass index will be measured.
* They will have a Cardio-Ankle Vascular Index (CAVI) test of the arteries. Blood pressure will be taken in the arms and legs and the heart will be monitored.
* Blood will be drawn. Participants will fast for 8 12 hours before this.
* Women will have a pregnancy test.
* Eligible participants will get a 2-week supply of niacin. They will take 2 tablets daily for one week, then 4 daily.
* Visit 2 will be 2 weeks after visit 1 and the niacin dose will be increased. Visit 3 will be 16 weeks after visit 1, and participants will stop taking niacin. Visit 4 will be 4 6 weeks after stopping niacin.
* During study visits, participants will repeat visit 1 tests.

DETAILED DESCRIPTION:
This single center clinical pilot study will investigate the effects of niacin on blood lipids and lipoprotein composition in human subjects who are healthy. Niacin (vitamin B3 or nicotinic acid) is a common nutrient found in many foods and is currently sold over the counter as a nutritional supplement. Extended-release versions of niacin are available over the counter (e.g., Slo-Niacin) or by prescription (Niaspan) and help to alleviate symptoms of flushing associated with larger doses of the vitamin. Studies of the effects of niacin therapy on clinical lipid measures consistently indicate a shift toward a healthier lipoprotein profile with increased HDL-C and decreases in both triglyceride and LDL-C. Despite this favorable shift in lipid profile, cardiovascular outcome studies on patients receiving niacin alone or in combination with statin therapy have resulted in mixed results creating uncertainty of the value of niacin therapy. The proposed study will examine in detail the effects of niacin therapy on lipoprotein composition and function, while also tracking measures of vascular health.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males and females who are at least 18 years of age at time of enrollment.
* Subject understands the investigational nature of the study and provides written, informed consent.

EXCLUSION CRITERIA:

* Subjects taking any lipid modification therapy, including but not limited to statins, fibrates and bile acid sequestrants.
* Subjects taking fish oil or any other supplements, which in the investigator s opinion may interfere with the study.
* Subjects with acute liver disease or active peptic ulcer disease.
* Subjects with elevated uric acid levels greater than 10 mg/dL or gout
* Pregnancy or women currently breastfeeding.
* Female subjects taking hormonal contraceptives or hormone replacement therapy may be included in this study only if they have been on a stable dose for at least 3 months.
* BMI less than 18.5
* Subjects with weight that varies greater than 20% over the past 3 months.
* Subjects taking the following medications for at least six weeks, which may interfere with the study, will be excluded: BAS, antibiotics, anticoagulants, anticonvulsants, antiarrhythmic, Cyclosporine, Mycophenolate and Synthroid. Subjects with chronic diarrhea, gastric bypass or lap band procedures, ostomies, bowel motility problems, or other conditions that could affect intestinal fat absorption.
* Subjects initiating new medications or patients on multiple medications may also be excluded.
* Inability to swallow capsules
* Patients with a history of type I or type II diabetes or HbA1c greater than 6.5%.
* Volunteers may also be excluded, if in the opinion of the study investigators, they have some other condition or disorder that may adversely affect the outcome of the study or the safety of the volunteer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0042.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function
Started | 22
Completed | 14
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in High-density Lipoprotein Protein Concentration
Description: Measure the mean percentage of niacin monotherapy on high-density lipoprotein (HDL) protein concentration
Time Frame: 20 weeks
Population: Out of the 14 participants that completed study, 3 participants were considered to be non-responders and not included in data analysis. Therefore, 11 participants were included in data analysis.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function
Number analyzed (Participants) | 11
Percentage Change
  High-density lipoprotein cholesterol | 16.0 (11.1)
  Low-density lipoprotein cholesterol | -20.0 (24.7)
  Triglyceride | -15.0 (21.2)
  Total Cholesterol | -11.0 (13.2)

2. Primary Outcome: Change in Proteins of High-density Lipoprotein Protein Composition on Niacin Monotherapy
Description: Measure the effect proteins with changes in protein composition of niacin monotherapy on high-density lipoprotein (HDL) protein composition. High-density lipoprotein protein were measured using Nuclear magnetic resonance (NMR) spectroscopy. NMR spectroscopy is a technique that uses the magnetic properties of atomic nuclei to analyze the chemical and physical properties of molecules or atoms. NMR spectroscopy is non-destructive and non-invasive, and can be used to study the structure, dynamics, and chemical reactions of molecules. NMR procedures numerical results which are comparable to laboratory results, and these data were used to measure the outcomes reported.
Time Frame: 20 weeks
Population: as for outcome 1
Measure: Number; unit: proteins
Units Other Than Participants: Proteins
Arm/Group | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function
Number analyzed (Participants) | 11
Number analyzed (Proteins) | 5
proteins | 5

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Adverse events were pre-specified to be collected as a single Arm/Group irrespective of dose level.
Arm/Group | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niacin ER in Healthy Participants and Its Effects on Lipoprotein Composition and Function (N=22)
Palpitations (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
CPK increased (Investigations) | 1
Low Thyroid Function (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02322203/Prot_SAP_000.pdf